CLINICAL TRIAL: NCT03083158
Title: Identification of Age-dependent Mechanism of Vaccine-induced Immunity to a Single Dose of Hepatitis B Vaccine Using a Systems Biology Approach - a Demonstration Project
Brief Title: Immunity to Hepatitis B Vaccine
Acronym: HVP01
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Vanderbilt University (Other); J. Craig Venter Institute (Other); The Scripps Research Institute (Other); University of California, San Diego (Other); Institut Pasteur (Industry); Human Vaccines Project (Other)
Responsible Party: Principal Investigator, Manish Sadarangani, Principle Investigator, University of British Columbia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: H17-00175
Record Dates: First submitted 2017-03-09; First posted 2017-03-17 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Hepatitis B; Immunization; Infection
MeSH Terms: conditions — Hepatitis B; Infections | interventions — Hepatitis B Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Other): Older adults, aged 61-80 years
  Interventions: Drug: Hepatitis B vaccine
- Group 2 (Other): Younger adults, aged 40-60 years
  Interventions: Drug: Hepatitis B vaccine

INTERVENTIONS:
Drug: Hepatitis B vaccine — 1.0 ml (20 micrograms) suspension of hepatitis B surface antigen for intramuscular injection
  Other Names: ENGERIX®-B

SUMMARY:
Infection and cancer is a major cause of death and morbidity, and may be preventable through vaccination. It is not fully understood at the molecular level why some people respond better than others to vaccines until now the technology to assess this has not been available. This has impaired vaccine development. The overall goal of the Human Vaccines Project is to understand the 'rules' of how vaccines work. In this demonstration project the investigators will vaccinate healthy adults with hepatitis B vaccine to start to understand better how it works, ultimately helping with rational vaccine design in the future.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult, corresponding to one of the study age groups.
* No history of hepatitis B disease.
* No prior receipt of any hepatitis B-containing vaccine.
* Undetectable level of anti-HBs and anti-HBc antibody and HBs antigen at study enrolment (indicating no evidence of prior hepatitis B vaccination or infection).
* Generally good health (stable chronic conditions acceptable), living independently or with minimal assistance (Clinical Frailty score 1-5) and able to attend clinic appointments.
* Willing and able to comply with the requirements of the protocol.
* Has given informed consent for participation in the study.

Exclusion Criteria:

The participant may not enter the study if ANY of the following apply:

* Individual who is on the delegation log for this study
* History of being a household contact of a known hepatitis B-infected individual.
* Planned administration of any vaccine not specified in the study protocol from 1 month pre- to the 1 month post-1st dose of vaccine.
* Planned receipt of any investigational drug for the duration of the study.
* Confirmed or suspected immunodeficiency.
* A family history of congenital or hereditary immunodeficiency.
* Receipt of more than 1 week of immunosuppressants or immune modifying drugs (e.g. oral prednisolone >0.5ml/kg/day or intravenous glucocorticoid steroid) in the 3 months prior to dose 1 of vaccine. Nasal, topical or inhaled steroids are allowed.
* Currently taking any anti-platelet or anti-coagulant medications (does not include daily low-dose aspirin).
* Bleeding disorder or thrombocytopenia, that contraindicates IM injection, blood collection and/or lymph node fine needle aspiration.
* Administration of immunoglobulins within the prior 12 months and/or any other blood products within the prior 3 months or planned during the study period.
* Current pregnancy or planning to become pregnant in the 6 months post-dose 1 vaccination.
* History of allergy to any component of the vaccine.
* Unstable medical condition, as indicated by a requirement for hospitalization or a substantial medication change to stabilize said condition within previous 3 months.
* History of any neurologic disorders or seizures, including a history of Guillain-Barre syndrome.
* Clinical Frailty score of 6-7 (moderately frail or severely frail).
* Scheduled elective surgery or other procedures requiring general anaesthesia from 1 month pre- to the 1 month post-1st dose of vaccine.
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.
* Temporary exclusion if acute symptomatic illness in the 7 days prior to planned first vaccine dose - vaccination will be delayed, but participant can remain in the study.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Antibody response to the first dose of hepatitis B vaccine | 28 days post-vaccination following the first dose of vaccine
  Anti-HBs antibody level

SECONDARY OUTCOMES:
Kinetics of the immune response to the first dose of hepatitis B vaccine with respect to cellular immune response | Baseline (pre-vaccine) and on days 1, 3, 7 and 14 post-vaccination
  Immunophenotyping by flow cytometric analysis of immune cell populations, including antigen-specific T-cell and B-cell responses, and response of immune cells to various stimuli in vitro
Kinetics of the immune response to the first dose of hepatitis B vaccine with respect to transcriptomic response | Baseline (pre-vaccine) and on days 1, 3, 7 and 14 post-vaccination
  Gene expression by RNA sequencing of whole blood and single immune cells
Kinetics of the immune response to the first dose of hepatitis B vaccine with respect to proteomic response | Baseline (pre-vaccine) and on days 1, 3, 7 and 14 post-vaccination
  Proteomic analysis of plasma and white blood cells
Kinetics of the immune response to the first dose of hepatitis B vaccine with respect to metabalomic response | Baseline (pre-vaccine) and on days 1, 3, 7 and 14 post-vaccination
  Metabolomic analysis of plasma
Kinetics of the immune response to the first dose of hepatitis B vaccine with respect to epigenetic response | Baseline (pre-vaccine) and on days 1, 3, 7 and 14 post-vaccination
  Epigenetic changes in genome
Kinetics of the immune response to the first dose of hepatitis B vaccine with respect to lymph node response | Pre-vaccine and 14 days following first dose only
  Immune responses in local lymph node, and comparison with peripheral blood responses
Identify the DNA sequence of B- and T- cell receptors following vaccination | Baseline (pre-vaccine) and on days 1, 3, 7 and 14 post-vaccination
  DNA sequencing of T- and B- cells

OTHER OUTCOMES:
To correlate the 'omics immune responses measured after the first dose with antibody level after the 1st and 3rd doses | Days 1, 3, 7 and 14 post-first dose of vaccine and 28 days after the 1st and 3rd doses of vaccine
  Correlation of immune endpoints (all secondary endpoints - outcomes 2 to 8) at days 1, 3, 7 and 14 post-first dose of vaccine and anti-HBs antibody level 28 days after the 1st and 3rd doses of vaccine
The influence of the gut, skin, buccal and nasal microbiota on responses to a single dose of hepatitis B vaccine - microbiome measured by 16S rDNA sequencing and vaccine response measured by anti-HBS antibody | Day 14 pre-first dose of vaccine and day 28 post-first dose of vaccine
  Correlation of gut, skin, buccal and nasal microbiota (obtained pre-vaccination) with HBV vaccine response.
The influence of a single dose of hepatitis B vaccine on the gut, skin, buccal and nasal microbiota - microbiome measured by 16S rDNA sequencing and vaccine response measured by anti-HBS antibody | Day 14 post-first dose of vaccine
  Analysis of changes in gut, skin, buccal and nasal microbiota obtained following vaccination
The quality of the antibody response following hepatitis B vaccination, measured by antibody subclass and avidity | Pre-vaccine and 1 month after the 1st dose, 5 months after the 2nd dose (6 months after 1st dose) and 1 month after the 3rd dose of vaccine
  Analysis of antibody subclass and avidity pre-vaccine and 1 month after the 1st dose, 5 months after the 2nd dose (6 months after 1st dose) and 1 month after the 3rd dose of vaccine
The genetic changes in B- and T-cells following doses of hepatitis B vaccine, measured by T cell and B cell receptpr sequencing | 28 days after the 1st dose, 7 days and 5 months after the 2nd dose (6 months after the 1st dose) and 7 days and 28 days after the 3rd dose of hepatitis B vaccine
  DNA sequencing of B- and T- cells 28 days after the 1st dose, 7 days and 5 months after the 2nd dose (6 months after the 1st dose) and 7 days and 28 days after the 3rd dose of hepatitis B vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Manish Sadarangani, Principal Investigator — University of British Columbia; Tobi Kollmann, Principal Investigator — University of British Columbia
Locations (1):
- Vaccine Evaluation Center, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — http://vaccineevaluationcenter.ca/